CLINICAL TRIAL: NCT00002472
Title: Phase II Pre-Irradiation Chemotherapy for Central Nervous System Germ Cell Malignancies
Brief Title: Cisplatin and Etoposide Prior to Radiation Therapy in Treating Patients With CNS Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jan C. Buckner , MD, Mayo Clinic
Purpose: Treatment
Other Study IDs: CDR0000076756; P30CA015083 (NIH); 891351 (Other: Mayo Clinic Cancer Center); T92-0208D (Other: NCI protocol)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Brain and Central Nervous System Tumors; Pediatric Germ Cell Tumor; Extragonadal Germ Cell Tumor
Keywords: childhood central nervous system germ cell tumor; extragonadal germ cell tumor; adult central nervous system germ cell tumor; childhood teratoma; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Teratoma | interventions — Cisplatin; Etoposide; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin and etoposide in treating patients with CNS tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with newly diagnosed CNS germ cell tumors treated with cisplatin and etoposide.
* Determine the survival of patients with CNS germ cell tumors treated with cisplatin and etoposide followed by cranial radiotherapy.
* Determine endocrine and cognitive function in these patients before and after receiving this regimen.

OUTLINE: Patients are stratified by histology (germinoma vs nongerminoma).

Patients receive cisplatin IV over 4 hours followed by etoposide IV over 30-60 minutes on days 1-5. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of 4 courses, patients with nongerminoma who achieve complete response (CR) and all patients with germinoma proceed to radiotherapy. After completion of 4 courses, patients with nongerminoma who achieve less than CR undergo resection of any residual cranial masses, if feasible, and then proceed to radiotherapy. Patients who experience disease progression or unacceptable toxicity during chemotherapy are restaged and proceed directly to radiotherapy.

Beginning a minimum of 3 weeks after completion of the last course of chemotherapy and after recovering from any toxic effects of chemotherapy, eligible patients undergo a regimen of craniospinal axis irradiation and/or localized cranial or spinal field irradiation based on histology, extent of disease, and response to chemotherapy. Patients with gross spinal meningeal disease after completion of chemotherapy undergo radiotherapy boost.

Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 12-25 patients with germinoma will be accrued for this study within 3-6 years. A total of 12-25 patients with nongerminoma will be accrued for this study within 6-12 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven CNS germ cell tumor of 1 of the following subtypes:

  * CNS germinoma
  * Immature teratoma
  * Embryonal cell carcinoma
  * Yolk sac tumor
  * Endodermal sinus tumor
  * Choriocarcinoma OR
* Pineal or suprasellar mass associated with elevated CSF alpha fetoprotein or beta-human chorionic gonadotropin allowed
* Patients 18 years and over with localized pure germinomas ineligible
* Evaluable CT or MRI of brain and/or spinal cord required

PATIENT CHARACTERISTICS:

Age:

* 3 and over

Hematopoietic:

* Age 18 and over:

  * WBC at least 4,000/mm^3
  * Platelet count at least 100,000/mm^3
* Under age 18:

  * Absolute neutrophil count at least 1,000/mm^3
  * Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 0.3 mg/dL above upper limit of normal for age

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for CNS germ cell tumor

Endocrine therapy:

* Concurrent corticosteroids allowed except as antiemetics

Radiotherapy:

* No prior cranial or spinal radiotherapy

Surgery:

* Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response rate
Survival
Endocrine and cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Jan C. Buckner, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota